CLINICAL TRIAL: NCT01475461
Title: A Phase 2, Randomized, Double-blinded, Placebo-controlled, Dose-ranging, Parallel Group Study To Evaluate Safety And Efficacy Of Pf-04937319 And Sitagliptin On Glycemic Control In Adult Patients With Type 2 Diabetes Mellitus Inadequately Controlled On Metformin
Brief Title: Phase 2 Study To Evaluate Safety And Efficacy Of Investigational Drug - PF04937319 In Patients With Type 2 Diabetes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: B1621007; 2011-004002-25 (EudraCT Number)
Record Dates: First submitted 2011-09-15; First posted 2011-11-21 (Estimated); Results first posted 2017-01-31 (Estimated); Last update posted 2017-01-31 (Estimated); Status verified 2016-12

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Phase 2; type 2 diabetes mellitus; PF-04937319
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — N,N-dimethyl-5-((2-methyl-6-((5-methylpyrazin-2-yl)carbamoyl)benzofuran-4-yl)oxy)pyrimidine-2-carboxamide; Sitagliptin Phosphate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- PF-04937319 - Dose 1 (Experimental)
  Interventions: Drug: PF-04937319 - 3mg
- PF-04937319 - Dose 2 (Experimental)
  Interventions: Drug: PF-04937319 - 20mg
- PF-04937319 - Dose 3 (Experimental)
  Interventions: Drug: PF-04937319 - 50mg
- PF-04937319 - Dose 4 (Experimental)
  Interventions: Drug: PF-04937319 - 100mg
- Sitagliptin (Active Comparator)
  Interventions: Drug: Sitagliptin - 100mg

INTERVENTIONS:
Drug: Placebo — double-dummy placebo tablets administered once-daily for 84-days
  Arms: Placebo
Drug: PF-04937319 - 3mg — PF-04937319 3mg administered as tablets once-daily for 84-days
  Arms: PF-04937319 - Dose 1
Drug: PF-04937319 - 20mg — PF-04937319 20mg administered as tablets once-daily for 84-days
  Arms: PF-04937319 - Dose 2
Drug: PF-04937319 - 50mg — PF-04937319 50mg administered as tablets once-daily for 84-days
  Arms: PF-04937319 - Dose 3
Drug: PF-04937319 - 100mg — PF-04937319 100mg administered as tablets once-daily for 84-days
  Arms: PF-04937319 - Dose 4
Drug: Sitagliptin - 100mg — Sitagliptin 100mg administered as tablets once-daily for 84-days
  Arms: Sitagliptin

SUMMARY:
B1621007 is designed to study the safety and efficacy of PF-04937319 in patients with type 2 diabetes

ELIGIBILITY:
Inclusion Criteria:

* patients with type 2 diabetes, on metformin, age between 18-55 yrs, male or female

Exclusion Criteria:

* patients with type 1 diabetes, medically unstable, unacceptable clinical laboratory test results at screening

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 345 (Actual)
Dates: Start 2011-11; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (62):
- United States (24):
  - Anaheim Clinical Trials, Anaheim, California
  - National Research Institute, Los Angeles, California
  - Encompass Clinical Research, Spring Valley, California
  - The Family Doctors of Belleview, Belleview, Florida
  - Swiss Medical Research, Miami, Florida
  - Renstar Medical Research, Ocala, Florida
  - Rockdale Medical Research Associates, Conyers, Georgia
  - Solaris Clinical Research, Meridian, Idaho
  - Central Kentucky Research Associates, Inc., Mount Sterling, Kentucky
  - Mount Sterling Clinic, Mount Sterling, Kentucky
  - The Office of Dr. Matthew S. Barton, MD, Las Vegas, Nevada
  - TKL Research, Inc., Paramus, New Jersey
  - Rochester Clinical Research, Inc., Rochester, New York
  - Lillestol Research, LLC, Fargo, North Dakota
  - PriMed Clinical Research, Kettering, Ohio
  - PriMed Physicians, Kettering, Ohio
  - Lynn Health Science Institute, Oklahoma City, Oklahoma
  - Medical Research South, LLC, Charleston, South Carolina
  - Newton Family Medicine, Charleston, South Carolina
  - Austin Center for Clinical Research, Austin, Texas
  - Texas Center for Drug Development, Inc., Houston, Texas
  - Plano Primary Care Clinic, Plano, Texas
  - Pioneer Research Solutions, Inc., Sugar Land, Texas
  - Martin Diagnostic Clinic, Tomball, Texas
- Hungary (9):
  - DRC Kft., Balatonfüred
  - Dr. Rethy Pal Korhaz-Rendelointezet, Békéscsaba
  - Qualiclinic Kft., Budapest
  - Debreceni Egyetem Orvos- es Egeszsegtudomanyi Centrum, Debrecen
  - Kenezy Korhaz Rendelointezet Egeszsegugyi Nonprofit Kft., Debrecen
  - Petz Aladar Megyei Oktato Korhaz, Győr
  - Polgar es Tersege Egeszsegugyi Kozpont Nonprofit Zrt., Polgár
  - Szegedi Tudomanyegyetem Szent-Gyorgyi Albert Klinikai Kozpont, Szeged
  - Zala Megyei Korhaz, Zalaegerszeg
- India (4):
  - Bhatia Hospital, Mumbai, Maharashtra
  - Seth G S Medical College & KEM Hospital, Dept of Endocrinology,, Mumbai, Maharashtra
  - Jehangir Clinical Development Centre Pvt. Ltd., Pune, Maharashtra
  - S.R. Kalla Memorial Gastro and General Hospital, Jaipur, Rajasthan
- Philippines (3):
  - Vicente Sotto Memorial Medical Center, Cebu City
  - Institute for Studies on Diabetes Foundation Inc., Marikina City
  - The Medical City, Pasig
- Romania (2):
  - Spitalul Clinic Judetean de Urgenta Cluj-Napoca, Cluj-Napoca, Jud. Cluj
  - Institutul National de Diabet, Nutritie si Boli Metabolice Prof. Dr. N. Paulescu, Bucharest
- Slovakia (8):
  - Metabolicke centrum MUDr. Katariny Raslovej, s.r.o., Bratislava
  - Medispektrum Plus, s.r.o., Bratislava
  - IN-DIA, s.r.o., Lučenec
  - MUDr. Zuzana Ochodnicka, Interna diabetologicka ambulancia, s.r.o., Nitra
  - NOEMIS, s.r.o., Nové Mesto nad Váhom
  - DIABETOL, s.r.o., Prešov
  - Areteus, s.r.o., Trebišov
  - Diabetes centrum, s.r.o., Trenčín
- South Africa (8):
  - Bloemfontein Medi-Clinic, Bloemfontein, Free State
  - Dr DR Lakha's Practice, Johannesburg, Gauteng
  - Midrand Medical Centre, Midrand, Gauteng
  - Medi-Clinic Heart Hospital, Pretoria, Gauteng
  - Dr Bhana, Waverley, Gauteng
  - Dr JH Mynhardt, Kimberley, Northern Cape
  - Randles Road Medical Centre, Durban
  - AA Mahomed Medical Centre, Moloto South
- Taiwan (4):
  - Changhua Christian Hospital, Changhua
  - Far Eastern Memorial Hospital, Division of Endocrinology and Metabolism, New Taipei City
  - Taichung Veterans General Hospital, Division of Metabolism and Endocrinology, Taichung
  - Chi Mei Medical Center, Tainan

REFERENCES:
- [Derived] Amin NB, Aggarwal N, Pall D, Paragh G, Denney WS, Le V, Riggs M, Calle RA. Two dose-ranging studies with PF-04937319, a systemic partial activator of glucokinase, as add-on therapy to metformin in adults with type 2 diabetes. Diabetes Obes Metab. 2015 Aug;17(8):751-9. doi: 10.1111/dom.12474. Epub 2015 May 11. PMID 25885172
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B1621007&StudyName=Phase%202%20Study%20To%20Evaluate%20Safety%20And%20Efficacy%20Of%20Investigational%20Drug%20-%20PF04937319%20In%20Patients%20With%20Type%202%20Diabetes

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Total 615 participants were consented,of which 376 participants entered to run-in period to receive sponsor provided Metformin, 345 participants then randomized to study treatment,of these 335 were treated. Results were collected for 335 participants as data from 1 site (10 participants) were excluded due to major good clinical practice violations.
Groups:
- Metformin 500 mg: Metformin 500 milligram (mg) immediate release tablet used as standardized, pre-specified background therapy in all participants initiated at the run-in visit and continued till follow-up visit.
- Placebo: Placebo matched to PF-04937319 tablet orally once daily and placebo matched to sitagliptin tablet orally once daily along with background metformin 500 mg immediate release tablets or as per standard clinical practice, for 12 weeks.
- PF-04937319 3 mg: PF-04937319 3 mg tablet orally once daily along with background metformin 500 mg immediate release tablets or as per standard clinical practice, for 12 weeks.
- PF-04937319 20 mg: PF-04937319 20 mg tablet orally once daily along with background metformin 500 mg immediate release tablets or as per standard clinical practice, for 12 weeks.
- PF-04937319 50 mg: PF-04937319 50 mg tablet orally once daily along with background metformin 500 mg immediate release tablets or as per standard clinical practice, for 12 weeks.
- PF-04937319 100 mg: PF-04937319 100 mg tablet orally once daily along with background metformin 500 mg immediate release tablets or as per standard clinical practice, for 12 weeks.
- Sitagliptin 100 mg: Sitagliptin 100 mg tablet orally once daily along with background metformin 500 mg immediate release tablets or as per standard clinical practice, for 12 weeks.
Period: Run-in Period
Arm/Group | Metformin 500 mg | Placebo | PF-04937319 3 mg | PF-04937319 20 mg | PF-04937319 50 mg | PF-04937319 100 mg | Sitagliptin 100 mg
Started | 376 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 335 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 41 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Not meet eligibility criteria | 16 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 7 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 11 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Other | 3 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 4 | 0 | 0 | 0 | 0 | 0 | 0
Period: Treatment Period
Arm/Group | Metformin 500 mg | Placebo | PF-04937319 3 mg | PF-04937319 20 mg | PF-04937319 50 mg | PF-04937319 100 mg | Sitagliptin 100 mg
Started | 0 | 57 | 57 | 54 | 56 | 56 | 55
Completed | 0 | 48 | 53 | 46 | 52 | 51 | 53
Not Completed | 0 | 9 | 4 | 8 | 4 | 5 | 2
Not completed — Death | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 3 | 2 | 3 | 1 | 2 | 1
Not completed — Withdrawal by Subject | 0 | 2 | 2 | 0 | 2 | 2 | 0
Not completed — Other | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 0 | 1 | 0 | 0 | 0 | 0 | 1
Not completed — Lack of Efficacy | 0 | 2 | 0 | 2 | 1 | 1 | 0
Not completed — Medication Error | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Baseline analysis population included all randomized participants who received at least 1 dose of study treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | PF-04937319 3 mg | PF-04937319 20 mg | PF-04937319 50 mg | PF-04937319 100 mg | Sitagliptin 100 mg | Total
Number analyzed (Participants) | 57 | 57 | 54 | 56 | 56 | 55 | 335
Age, Customized [Number; unit: Participants]
  >=18 to =<44 years | 15 | 17 | 14 | 15 | 15 | 17 | 93
  >=45 to =<64 years | 42 | 40 | 40 | 41 | 41 | 38 | 242
Gender [Count of Participants; unit: Participants]
  Female | 21 | 29 | 22 | 23 | 26 | 22 | 143
  Male | 36 | 28 | 32 | 33 | 30 | 33 | 192

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Glycosylated Hemoglobin (HbA1C) at Week 12
Description: HbA1c is a form of hemoglobin which is measured primarily to identify the average glycemic control over prolonged periods of time. The normal range for the HbA1c test, was identified as less than (<) 6.5 percent (%) by the study-specific central laboratory used. Change from baseline in percentage of HbA1c in participants were reported.
Time Frame: Baseline (Day 1), Week 12
Population: Full analysis set (FAS) included all randomized participants who received at least 1 dose of study treatment. Here, 'N' (number of participants analyzed) signifies participants for whom data was summarized for this measure and 'n' signifies participants evaluable at given time points for each group.
Measure: Mean (Standard Deviation); unit: percentage of hemoglobin
Groups:
- Placebo: Placebo matched to PF-04937319 tablet orally once daily and placebo matched to sitagliptin tablet orally once daily along with background metformin 500 milligram (mg) immediate release tablets or as per standard clinical practice, for 12 weeks.
- PF-04937319 3 mg: PF-04937319 3 mg tablet orally once daily along with background metformin 500 milligram (mg) immediate release tablets or as per standard clinical practice, for 12 weeks.
- PF-04937319 20 mg: PF-04937319 20 mg tablet orally once daily along with background metformin 500 milligram (mg) immediate release tablets or as per standard clinical practice, for 12 weeks.
- PF-04937319 50 mg: PF-04937319 50 mg tablet orally once daily along with background metformin 500 milligram (mg) immediate release tablets or as per standard clinical practice, for 12 weeks.
- PF-04937319 100 mg: PF-04937319 100 mg tablet orally once daily along with background metformin 500 milligram (mg) immediate release tablets or as per standard clinical practice, for 12 weeks.
- Sitagliptin: Sitagliptin 100 mg tablet orally once daily along with background metformin 500 milligram (mg) immediate release tablets or as per standard clinical practice, for 12 weeks.
Arm/Group | Placebo | PF-04937319 3 mg | PF-04937319 20 mg | PF-04937319 50 mg | PF-04937319 100 mg | Sitagliptin
Number analyzed (Participants) | 50 | 55 | 48 | 55 | 53 | 53
percentage of hemoglobin
  Baseline (n=50,55,48,55,53,53) | 8.01 (1.099) | 8.00 (1.031) | 7.80 (0.965) | 8.15 (1.002) | 8.31 (1.043) | 7.89 (1.022)
  Change at Week 12 (n=46,52,45,52,50,53) | -0.42 (0.821) | -0.33 (0.793) | -0.53 (0.919) | -0.59 (0.988) | -0.80 (0.955) | -0.79 (0.859)
Statistical Analysis 1: Comparison: Placebo vs PF-04937319 3 mg; Week 12: Treatment difference and 80 percent(%) confidence interval (CI) were based on least squares (LS) mean. A mixed model repeated measure (MMRM) analysis was performed with treatment, time and treatment-by-time interaction as fixed effects, baseline as the covariate, time was repeated for participant. Null hypothesis stated there was no difference between PF 04937319 and placebo, alternative hypothesis stated PF 04937319 was superior to placebo; Test type: Superiority or Other; p = 0.5206, t-test, 1 sided — p-value was 1-sided; No adjustments were made for multiple comparisons among treatment groups; Least squares (LS) Mean Difference = 0.01, 80% CI 2-sided [-0.21 to 0.23], Standard Error of Mean 0.172
Statistical Analysis 2: Comparison: Placebo vs PF-04937319 20 mg; Week 12: Treatment difference and 80% CI were based on LS mean. MMRM analysis was performed with treatment, time and treatment-by-time interaction as fixed effects, baseline as the covariate, time was repeated for participant. Null hypothesis stated there was no difference between PF 04937319 and placebo, alternative hypothesis stated PF 04937319 was superior to placebo; Test type: Superiority or Other; p = 0.1645, t-test, 1 sided — p-value was 1-sided; No adjustments were made for multiple comparisons among treatment groups; LS Mean Difference = -0.17, 80% CI 2-sided [-0.40 to 0.05], Standard Error of Mean 0.178
Statistical Analysis 3: Comparison: Placebo vs PF-04937319 50 mg; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.1592, t-test, 1 sided — p-value was 1-sided; No adjustments were made for multiple comparisons among treatment groups; LS Mean Difference = -0.17, 80% CI 2-sided [-0.39 to 0.05], Standard Error of Mean 0.172
Statistical Analysis 4: Comparison: Placebo vs PF-04937319 100 mg; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.0049, t-test, 1 sided — p-value was 1-sided; LS Mean Difference = -0.45, 80% CI 2-sided [-0.68 to -0.23], Standard Error of Mean 0.174
Statistical Analysis 5: Comparison: Placebo vs Sitagliptin; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.0068, t-test, 1 sided — p-value was 1-sided; LS Mean Difference = -0.43, 80% CI 2-sided [-0.65 to -0.21], Standard Error of Mean 0.173

2. Secondary Outcome: Change From Baseline in Glycosylated Hemoglobin (HbA1C) at Week 2, 4 and 8
Description: HbA1c is a form of hemoglobin which is measured primarily to identify the average glycemic control over prolonged periods of time. The normal range for the HbA1c test, was identified as <6.5 percent by the study-specific central laboratory used. Change from baseline in percentage of HbA1c in participants were reported.
Time Frame: Baseline(Day 1), Week 2, 4, 8
Population: FAS: All randomized participants who received at least 1 dose of study treatment. Here, 'N' signifies participants for whom data was summarized for this measure and 'n' signifies participants who were evaluable at given time points for each group. Data for Week 2 had not been reported because as per protocol it was not intended to be collected.
Measure: Mean (Standard Deviation); unit: percentage of hemoglobin
Arm/Group | Placebo | PF-04937319 3 mg | PF-04937319 20 mg | PF-04937319 50 mg | PF-04937319 100 mg | Sitagliptin
Number analyzed (Participants) | 50 | 55 | 48 | 55 | 53 | 53
percentage of hemoglobin
  Change at Week 4 (n= 50, 55, 48, 55, 53, 53) | -0.20 (0.397) | -0.24 (0.568) | -0.32 (0.520) | -0.35 (0.601) | -0.50 (0.470) | -0.52 (0.503)
  Change at Week 8 (n=48, 53, 45, 52, 50, 51) | -0.36 (0.664) | -0.32 (0.781) | -0.46 (0.803) | -0.50 (0.848) | -0.86 (0.726) | -0.77 (0.699)
Statistical Analysis 1: Comparison: Placebo vs PF-04937319 3 mg; Week 4: Treatment difference and 80 percent(%) confidence interval (CI) were based on least squares (LS) mean. A mixed model repeated measure (MMRM) analysis was performed with treatment, time and treatment-by-time interaction as fixed effects, baseline as the covariate, time was repeated for participant; Test type: Superiority or Other; p = 0.3434, t-test, 1 sided — p-value was 1-sided; LS Mean Difference = -0.04, 80% CI 2-sided [-0.16 to 0.09], Standard Error of Mean 0.097
Statistical Analysis 2: Comparison: Placebo vs PF-04937319 20 mg; Week 4: Treatment difference and 80% CI were based on LS mean. MMRM analysis was performed with treatment, time and treatment-by-time interaction as fixed effects, baseline, as the covariates, time was repeated for participant; Test type: Superiority or Other; p = 0.0892, t-test, 1 sided — p-value was 1-sided; LS Mean Difference = -0.14, 80% CI 2-sided [-0.27 to -0.01], Standard Error of Mean 0.101
Statistical Analysis 3: Comparison: Placebo vs PF-04937319 50 mg; [analysis description as in outcome 2, analysis 2]; Test type: Superiority or Other; p = 0.0826, t-test, 1 sided — p-value was 1-sided; LS Mean Difference = -0.14, 80% CI 2-sided [-0.26 to -0.01], Standard Error of Mean 0.097
Statistical Analysis 4: Comparison: Placebo vs PF-04937319 100 mg; [analysis description as in outcome 2, analysis 2]; Test type: Superiority or Other; p = 0.0031, t-test, 1 sided — p-value was 1-sided; LS Mean Difference = -0.27, 80% CI 2-sided [-0.40 to -0.15], Standard Error of Mean 0.098
Statistical Analysis 5: Comparison: Placebo vs Sitagliptin; Week 4: Treatment difference and 80% CI were based on LS mean. MMRM analysis was performed with treatment, time and treatment-by-time interaction as fixed effects, baseline as the covariate, time was repeated for participant; Test type: Superiority or Other; p = 0.0005, t-test, 1 sided — p-value was 1-sided; LS Mean Difference = -0.33, 80% CI 2-sided [-0.45 to -0.20], Standard Error of Mean 0.098
Statistical Analysis 6: Comparison: Placebo vs PF-04937319 3 mg; Week 8: Treatment difference and 80% CI were based on LS mean. MMRM analysis was performed with treatment, time and treatment-by-time interaction as fixed effects, baseline as the covariate, time was repeated for participant; Test type: Superiority or Other; p = 0.5133, t-test, 1 sided — p-value was 1-sided; LS Mean Difference = 0.00, 80% CI 2-sided [-0.18 to 0.19], Standard Error of Mean 0.144
Statistical Analysis 7: Comparison: Placebo vs PF-04937319 20 mg; [analysis description as in outcome 2, analysis 6]; Test type: Superiority or Other; p = 0.1873, t-test, 1 sided — p-value was 1-sided; LS Mean Difference = -0.13, 80% CI 2-sided [-0.33 to 0.06], Standard Error of Mean 0.150
Statistical Analysis 8: Comparison: Placebo vs PF-04937319 50 mg; [analysis description as in outcome 2, analysis 6]; Test type: Superiority or Other; p = 0.2120, t-test, 1 sided — p-value was 1-sided; LS Mean Difference = -0.12, 80% CI 2-sided [-0.30 to 0.07], Standard Error of Mean 0.145
Statistical Analysis 9: Comparison: Placebo vs PF-04937319 100 mg; Week 8: Treatment difference and 80% CI were based on LS mean. MMRM analysis was performed with treatment, time and treatment-by-time interaction as fixed effects, baseline, as the covariates, time was repeated for participant; Test type: Superiority or Other; p = 0.0001, t-test, 1 sided — p-value was 1-sided; LS Mean Difference = -0.54, 80% CI 2-sided [-0.73 to -0.35], Standard Error of Mean 0.146
Statistical Analysis 10: Comparison: Placebo vs Sitagliptin; [analysis description as in outcome 2, analysis 6]; Test type: Superiority or Other; p = 0.0021, t-test, 1 sided — p-value was 1-sided; LS Mean Difference = -0.42, 80% CI 2-sided [-0.61 to -0.23], Standard Error of Mean 0.146

3. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose at Week 1, 2, 4, 8, 12 and 14
Time Frame: Baseline (Day 1), Week 1, 2, 4, 8, 12, 14
Population: FAS: All randomized participants who received at least 1 dose of study treatment. Here, 'N' signifies participants for whom data was summarized for this measure and 'n' signifies participants who were evaluable at given time points for each group. Data for Week 1 had not been reported because as per protocol it was not intended to be collected.
Measure: Mean (Standard Deviation); unit: milligram per deciliter (mg/dL)
Arm/Group | Placebo | PF-04937319 3 mg | PF-04937319 20 mg | PF-04937319 50 mg | PF-04937319 100 mg | Sitagliptin
Number analyzed (Participants) | 56 | 56 | 52 | 56 | 55 | 55
milligram per deciliter (mg/dL)
  Baseline (n=56, 56, 52, 56, 55, 55) | 168.3 (42.99) | 159.8 (40.43) | 155.1 (37.74) | 166.1 (42.56) | 164.8 (41.14) | 160.7 (35.87)
  Change at Week 2 (n=54, 56, 50, 56, 54, 55) | -5.2 (26.22) | 0.7 (26.21) | -3.2 (19.67) | -6.8 (32.84) | -10.8 (25.73) | -13.6 (23.75)
  Change at Week 4 (n=52, 56, 51, 55, 54, 53) | -1.8 (31.25) | -0.3 (23.21) | -0.2 (21.29) | -8.3 (34.02) | -9.6 (29.30) | -19.3 (26.33)
  Change at Week 8 (n=50, 54, 47, 52, 51, 52) | -3.1 (37.03) | 0.7 (26.83) | -2.5 (27.49) | -15.2 (32.29) | -6.5 (29.50) | -15.4 (25.98)
  Change at Week 12 (n=48, 53, 47, 52, 51, 53) | -7.5 (31.21) | -2.5 (28.58) | -3.8 (31.62) | -10.8 (37.51) | 3.5 (41.74) | -12.9 (31.97)
  Change at Week 14 (n=45, 53, 46, 52, 51, 53) | -5.9 (33.18) | -3.5 (28.43) | -3.1 (32.62) | -1.0 (34.37) | 10.2 (38.62) | -2.6 (36.41)
Statistical Analysis 1: Comparison: Placebo vs PF-04937319 3 mg; Week 2: Treatment difference and 80 percent(%) confidence interval (CI) were based on least squares (LS) mean. A mixed model repeated measure (MMRM) analysis was performed with treatment, time and treatment-by-time interaction as fixed effects, baseline as the covariate, time was repeated for participant; Test type: Superiority or Other; p = 0.7240, t-test, 1 sided — p-value was 1-sided; LS Mean Difference = 2.87, 80% CI 2-sided [-3.32 to 9.07], Standard Error of Mean 4.823
Statistical Analysis 2: Comparison: Placebo vs PF-04937319 20 mg; Week 2: Treatment difference and 80% CI were based on LS mean. MMRM analysis was performed with treatment, time and treatment-by-time interaction as fixed effects, baseline as the covariate, time was repeated for participant; Test type: Superiority or Other; p = 0.3608, t-test, 1 sided — p-value was 1-sided; LS Mean Difference = -1.77, 80% CI 2-sided [-8.13 to 4.59], Standard Error of Mean 4.952
Statistical Analysis 3: Comparison: Placebo vs PF-04937319 50 mg; [analysis description as in outcome 3, analysis 2]; Test type: Superiority or Other; p = 0.2511, t-test, 1 sided — p-value was 1-sided; LS Mean Difference = -3.24, 80% CI 2-sided [-9.42 to 2.95], Standard Error of Mean 4.816
Statistical Analysis 4: Comparison: Placebo vs PF-04937319 100 mg; [analysis description as in outcome 3, analysis 2]; Test type: Superiority or Other; p = 0.0673, t-test, 1 sided — p-value was 1-sided; LS Mean Difference = -7.28, 80% CI 2-sided [-13.51 to -1.05], Standard Error of Mean 4.851
Statistical Analysis 5: Comparison: Placebo vs Sitagliptin; [analysis description as in outcome 3, analysis 2]; Test type: Superiority or Other; p = 0.0106, t-test, 1 sided — p-value was 1-sided; LS Mean Difference = -11.22, 80% CI 2-sided [-17.44 to -5.00], Standard Error of Mean 4.843
Statistical Analysis 6: Comparison: Placebo vs PF-04937319 3 mg; [analysis description as in outcome 2, analysis 5]; Test type: Superiority or Other; p = 0.4127, t-test, 1 sided — p-value was 1-sided; LS Mean Difference = -1.13, 80% CI 2-sided [-7.73 to 5.47], Standard Error of Mean 5.138
Statistical Analysis 7: Comparison: Placebo vs PF-04937319 20 mg; [analysis description as in outcome 2, analysis 5]; Test type: Superiority or Other; p = 0.3604, t-test, 1 sided — p-value was 1-sided; LS Mean Difference = -1.88, 80% CI 2-sided [-8.64 to 4.87], Standard Error of Mean 5.261
Statistical Analysis 8: Comparison: Placebo vs PF-04937319 50 mg; [analysis description as in outcome 2, analysis 5]; Test type: Superiority or Other; p = 0.0770, t-test, 1 sided — p-value was 1-sided; LS Mean Difference = -7.35, 80% CI 2-sided [-13.96 to -0.74], Standard Error of Mean 5.147
Statistical Analysis 9: Comparison: Placebo vs PF-04937319 100 mg; [analysis description as in outcome 2, analysis 5]; Test type: Superiority or Other; p = 0.0451, t-test, 1 sided — p-value was 1-sided; LS Mean Difference = -8.79, 80% CI 2-sided [-15.43 to -2.15], Standard Error of Mean 5.171
Statistical Analysis 10: Comparison: Placebo vs Sitagliptin; [analysis description as in outcome 2, analysis 5]; Test type: Superiority or Other; p = 0.0001, t-test, 1 sided — p-value was 1-sided; LS Mean Difference = -19.90, 80% CI 2-sided [-26.57 to -13.23], Standard Error of Mean 5.191
Statistical Analysis 11: Comparison: Placebo vs PF-04937319 3 mg; [analysis description as in outcome 2, analysis 6]; Test type: Superiority or Other; p = 0.5783, t-test, 1 sided — p-value was 1-sided; LS Mean Difference = 1.11, 80% CI 2-sided [-6.08 to 8.30], Standard Error of Mean 5.599
Statistical Analysis 12: Comparison: Placebo vs PF-04937319 20 mg; [analysis description as in outcome 2, analysis 6]; Test type: Superiority or Other; p = 0.3604, t-test, 1 sided — p-value was 1-sided; LS Mean Difference = -2.07, 80% CI 2-sided [-9.50 to 5.36], Standard Error of Mean 5.785
Statistical Analysis 13: Comparison: Placebo vs PF-04937319 50 mg; [analysis description as in outcome 2, analysis 6]; Test type: Superiority or Other; p = 0.0161, t-test, 1 sided — p-value was 1-sided; LS Mean Difference = -12.12, 80% CI 2-sided [-19.36 to -4.88], Standard Error of Mean 5.636
Statistical Analysis 14: Comparison: Placebo vs PF-04937319 100 mg; [analysis description as in outcome 2, analysis 6]; Test type: Superiority or Other; p = 0.2185, t-test, 1 sided — p-value was 1-sided; LS Mean Difference = -4.41, 80% CI 2-sided [-11.68 to 2.87], Standard Error of Mean 5.663
Statistical Analysis 15: Comparison: Placebo vs Sitagliptin; [analysis description as in outcome 2, analysis 6]; Test type: Superiority or Other; p = 0.0034, t-test, 1 sided — p-value was 1-sided; LS Mean Difference = -15.41, 80% CI 2-sided [-22.67 to -8.16], Standard Error of Mean 5.649
Statistical Analysis 16: Comparison: Placebo vs PF-04937319 3 mg; Week 12: Treatment difference and 80% CI were based on LS mean. MMRM analysis was performed with treatment, time and treatment-by-time interaction as fixed effects, baseline as the covariate, time was repeated for participant; Test type: Superiority or Other; p = 0.5727, t-test, 1 sided — p-value was 1-sided; LS Mean Difference = 1.17, 80% CI 2-sided [-7.03 to 9.37], Standard Error of Mean 6.387
Statistical Analysis 17: Comparison: Placebo vs PF-04937319 20 mg; [analysis description as in outcome 3, analysis 16]; Test type: Superiority or Other; p = 0.4961, t-test, 1 sided — p-value was 1-sided; LS Mean Difference = -0.06, 80% CI 2-sided [-8.51 to 8.38], Standard Error of Mean 6.578
Statistical Analysis 18: Comparison: Placebo vs PF-04937319 50 mg; [analysis description as in outcome 3, analysis 16]; Test type: Superiority or Other; p = 0.2616, t-test, 1 sided — p-value was 1-sided; LS Mean Difference = -4.10, 80% CI 2-sided [-12.33 to 4.14], Standard Error of Mean 6.411
Statistical Analysis 19: Comparison: Placebo vs PF-04937319 100 mg; [analysis description as in outcome 3, analysis 16]; Test type: Superiority or Other; p = 0.9197, t-test, 1 sided — p-value was 1-sided; LS Mean Difference = 9.06, 80% CI 2-sided [0.79 to 17.34], Standard Error of Mean 6.441
Statistical Analysis 20: Comparison: Placebo vs Sitagliptin; [analysis description as in outcome 3, analysis 16]; Test type: Superiority or Other; p = 0.0860, t-test, 1 sided — p-value was 1-sided; LS Mean Difference = -8.76, 80% CI 2-sided [-16.98 to -0.54], Standard Error of Mean 6.398
Statistical Analysis 21: Comparison: Placebo vs PF-04937319 3 mg; Week 14: Treatment difference and 80% CI were based on LS mean. MMRM analysis was performed with treatment, time and treatment-by-time interaction as fixed effects, baseline as the covariate, time was repeated for participant; Test type: Superiority or Other; p = 0.5132, t-test, 1 sided — p-value was 1-sided; LS Mean Difference = 0.22, 80% CI 2-sided [-8.10 to 8.53], Standard Error of Mean 6.476
Statistical Analysis 22: Comparison: Placebo vs PF-04937319 20 mg; [analysis description as in outcome 3, analysis 21]; Test type: Superiority or Other; p = 0.6560, t-test, 1 sided — p-value was 1-sided; LS Mean Difference = 2.68, 80% CI 2-sided [-5.89 to 11.26], Standard Error of Mean 6.676
Statistical Analysis 23: Comparison: Placebo vs PF-04937319 50 mg; [analysis description as in outcome 3, analysis 21]; Test type: Superiority or Other; p = 0.8285, t-test, 1 sided — p-value was 1-sided; LS Mean Difference = 6.17, 80% CI 2-sided [-2.17 to 14.52], Standard Error of Mean 6.496
Statistical Analysis 24: Comparison: Placebo vs PF-04937319 100 mg; [analysis description as in outcome 3, analysis 21]; Test type: Superiority or Other; p = 0.9925, t-test, 1 sided — p-value was 1-sided; LS Mean Difference = 15.98, 80% CI 2-sided [7.59 to 24.36], Standard Error of Mean 6.527
Statistical Analysis 25: Comparison: Placebo vs Sitagliptin; [analysis description as in outcome 3, analysis 21]; Test type: Superiority or Other; p = 0.6010, t-test, 1 sided — p-value was 1-sided; LS Mean Difference = 1.66, 80% CI 2-sided [-6.67 to 10.00], Standard Error of Mean 6.487

4. Secondary Outcome: Percentage of Participants Achieving Less Than 6.5 Percent and Less Than 7 Percent Glycosylated Hemoglobin (HbA1c) Levels at Week 12
Description: HbA1c is a form of hemoglobin which is measured primarily to identify the average glycemic control over prolonged periods of time. The normal range for the HbA1c test, was identified as <6.5 percent by the study-specific central laboratory used and data are presented in categories of <6.5 percent and <7 percent.
Time Frame: Week 12
Population: FAS: All randomized participants who received at least 1 dose of study treatment. Here, 'N' signifies participants for whom data was summarized for this measure.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | PF-04937319 3 mg | PF-04937319 20 mg | PF-04937319 50 mg | PF-04937319 100 mg | Sitagliptin
Number analyzed (Participants) | 48 | 53 | 47 | 52 | 51 | 53
percentage of participants
  <6.5 percent | 12.5 | 9.4 | 19.1 | 15.4 | 17.6 | 32.1
  <7 percent | 22.9 | 26.4 | 42.6 | 30.8 | 39.2 | 56.6

5. Secondary Outcome: Number of Participants With Increase From Baseline Electrocardiogram (ECG)Data
Description: Criteria for increase from baseline data: PR interval (percent change of greater than or equal to [>=] 25/50% [if baseline>200 then percent change of >25% counts; if baseline <=200 then percent change of >50% counts]; QRS complex (percent change of >=50%); QT Fridericia's correction (QTcF) interval (change of >=30 to <60 millisecond [msec], and change of >=60 msec).
Time Frame: Baseline (Day 1) up to Week 14
Population: Safety analysis set included all randomized participants who received at least 1 dose of study treatment. Here, 'N' signifies participants for whom data was collected for this measure.
Measure: Number; unit: participants
Arm/Group | Placebo | PF-04937319 3 mg | PF-04937319 20 mg | PF-04937319 50 mg | PF-04937319 100 mg | Sitagliptin
Number analyzed (Participants) | 53 | 57 | 52 | 56 | 55 | 54
participants
  PR interval: Percent change of >=25/50% | 0 | 1 | 0 | 0 | 1 | 2
  QRS interval: Percent change of >=50% | 0 | 1 | 1 | 1 | 1 | 1
  QTcF interval: Change of >=30 to <60 msec | 7 | 5 | 3 | 3 | 3 | 7
  QTcF interval: Change of >=60 msec | 1 | 0 | 0 | 1 | 2 | 0

6. Secondary Outcome: Number of Participants With Increase/Decrease From Baseline Vital Signs Data
Description: Participants who met the criteria for increase or decrease in vital signs data were reported. Criteria for increase or decrease from baseline vital signs data: sitting systolic blood pressure (BP) of >=30 millimeter of mercury (mmHg); sitting diastolic BP of >=20 mmHg and pulse rate was based on investigator's discretion.
Time Frame: Baseline (Day 1) up to Week 14
Population: as for outcome 5
Measure: Number; unit: participants
Arm/Group | Placebo | PF-04937319 3 mg | PF-04937319 20 mg | PF-04937319 50 mg | PF-04937319 100 mg | Sitagliptin
Number analyzed (Participants) | 56 | 57 | 53 | 56 | 55 | 55
participants
  Increase in systolic BP (>=30 mmHg) | 1 | 2 | 2 | 1 | 3 | 2
  Increase in diastolic BP (>=20 mmHg) | 1 | 4 | 0 | 1 | 4 | 2
  Decrease in systolic BP (>=30 mmHg) | 1 | 2 | 1 | 1 | 2 | 1
  Decrease in diastolic BP (>=20 mmHg) | 2 | 1 | 6 | 1 | 3 | 1

7. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (AEs) or Serious Adverse Events (SAEs)
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. An SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent are events between first dose of study drug and up to 14 days after last dose that were absent before treatment or that worsened relative to pretreatment state. AEs included both serious and non-serious adverse events.
Time Frame: Baseline (Day 1) up to 14 days after last dose (up to 101 days)
Population: Safety analysis set included all randomized participants who received at least 1 dose of study treatment.
Measure: Number; unit: participants
Groups:
- Sitagliptin 100 mg: Sitagliptin 100 mg tablet orally tablet once daily along with background metformin 500 mg immediate release tablets or as per standard clinical practice, for 12 weeks.
Arm/Group | Metformin 500 mg | Placebo | PF-04937319 3 mg | PF-04937319 20 mg | PF-04937319 50 mg | PF-04937319 100 mg | Sitagliptin 100 mg
Number analyzed (Participants) | 376 | 57 | 57 | 54 | 56 | 56 | 55
participants
  AEs | 37 | 19 | 19 | 19 | 16 | 24 | 18
  SAEs | 0 | 1 | 0 | 1 | 0 | 1 | 0

8. Secondary Outcome: Percentage of Participants With at Least 1 Hypoglycemic Events (HAE) Episode
Description: A hypoglycemic event (HAE) was identified by characteristic symptoms or blood glucose levels. HAE is defined as 1 of the given definitions: Characteristic symptoms of HAE with no home glucose monitoring performed where clinical picture included prompt resolution with food intake, subcutaneous glucagon, or intravenous glucose; or characteristic symptoms of HAE with home glucose monitoring measurement =< 70 milligram per deciliter (mg/dL) using ACCU-CHEK plasma-referenced home glucometers or =<74 mg/dL using International Federation of Clinical Chemistry (IFCC) referenced ACCU-CHEK or central laboratory glucometers; or any laboratory glucose value, meeting the following criterion with or without accompanying symptoms: =<49 mg/dL using ACCU-CHEK plasma-referenced home glucometers or =<53 mg/dL using IFCC referenced ACCU-CHEK or central laboratory glucometers.
Time Frame: Baseline (Day 1) up to Week 14
Population: as for outcome 5
Measure: Number; unit: percentage of participants
Arm/Group | Metformin 500 mg | Placebo | PF-04937319 3 mg | PF-04937319 20 mg | PF-04937319 50 mg | PF-04937319 100 mg | Sitagliptin 100 mg
Number analyzed (Participants) | 376 | 57 | 57 | 54 | 56 | 56 | 55
percentage of participants | 0 | 0 | 0 | 1 | 0 | 2 | 1

9. Secondary Outcome: Number of Hypoglycemic Events (HAE) Episodes Per Participant
Description: A hypoglycemic event (HAE) was identified by characteristic symptoms or blood glucose levels. Median number of events per participant was reported
Time Frame: Baseline (Day 1) up to Week 14
Population: as for outcome 5
Measure: Median (Full Range); unit: events per participant
Groups:
- Sitagliptin 100 mg: Sitagliptin 100 mg tablet orally once daily along with background metformin 500 milligram (mg) immediate release tablets or as per standard clinical practice, for 12 weeks.
Arm/Group | Metformin 500 mg | Placebo | PF-04937319 3 mg | PF-04937319 20 mg | PF-04937319 50 mg | PF-04937319 100 mg | Sitagliptin 100 mg
Number analyzed (Participants) | 376 | 57 | 57 | 54 | 56 | 56 | 56
events per participant | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 2] | 0 [0 to 0] | 0 [0 to 1] | 0 [0 to 2]

10. Secondary Outcome: Change From Baseline in Body Weight at Week 2, 4, 8, 12 and 14
Time Frame: Baseline (Day 1), Week 2, 4, 8 , 12 , 14
Population: Safety analysis set included all randomized participants who received at least 1 dose of study treatment. Here, 'N' signifies participants for whom data was collected for this measure and n=participants who were evaluable at given time points for each group.
Measure: Mean (Standard Deviation); unit: kilogram (kg)
Arm/Group | Placebo | PF-04937319 3 mg | PF-04937319 20 mg | PF-04937319 50 mg | PF-04937319 100 mg | Sitagliptin 100 mg
Number analyzed (Participants) | 55 | 55 | 50 | 56 | 54 | 55
kilogram (kg)
  Baseline (n=55, 55, 50, 56, 54, 55) | 86.446 (19.1859) | 87.865 (23.7732) | 88.371 (17.3923) | 88.066 (20.3446) | 91.239 (21.2731) | 87.025 (21.2567)
  Change at Week 2 (n=54, 55, 49, 56, 53, 55) | -0.239 (0.7264) | 0.435 (5.2348) | -0.052 (1.0570) | -0.283 (1.0520) | -0.053 (0.9010) | -0.384 (1.1041)
  Change at Week 4 (n=51, 55, 49, 55, 53, 53) | -0.704 (1.5651) | 0.214 (5.1426) | -0.192 (1.4649) | -0.203 (1.7609) | -0.374 (1.2083) | -0.353 (1.1598)
  Change at Week 8 (n=49, 53, 45, 52, 50, 52) | -0.823 (1.6750) | -0.003 (5.0869) | -0.510 (1.7467) | -0.270 (1.6559) | -0.475 (1.4374) | -0.702 (1.6095)
  Change at Week 12 (n=47, 52, 45, 52, 50, 53) | -0.804 (2.0119) | -0.142 (4.8928) | -0.455 (1.9213) | -0.352 (1.8121) | -0.623 (1.9647) | -0.917 (1.9591)
  Change at Week 14 (n=44, 52, 44, 52, 50, 53) | -0.588 (2.0994) | 0.011 (0.6634) | -0.613 (0.3149) | -0.492 (0.2823) | -0.916 (0.3743) | -1.172 (0.2850)
Statistical Analysis 1: Comparison: Placebo vs PF-04937319 3 mg; Week 2: Treatment difference and 80 percent (%) confidence interval (CI) were based on least squares (LS) mean. A mixed model repeated measure (MMRM) analysis was performed with treatment, time and treatment-by-time interaction as fixed effects, baseline as the covariate, time was repeated for participant; Test type: Superiority or Other; p = 0.0913, t-test, 2 sided — P-value was 2-sided; LS Mean Difference = 0.76, 80% CI 2-sided [0.18 to 1.34], Standard Error of Mean 0.449
Statistical Analysis 2: Comparison: Placebo vs PF-04937319 20 mg; [analysis description as in outcome 3, analysis 2]; Test type: Superiority or Other; p = 0.5236, t-test, 2 sided — P-value was 2-sided; LS Mean Difference = 0.29, 80% CI 2-sided [-0.30 to 0.89], Standard Error of Mean 0.461
Statistical Analysis 3: Comparison: Placebo vs PF-04937319 50 mg; [analysis description as in outcome 3, analysis 2]; Test type: Superiority or Other; p = 0.9244, t-test, 2 sided — P-value was 2-sided; LS Mean Difference = 0.04, 80% CI 2-sided [-0.53 to 0.62], Standard Error of Mean 0.447
Statistical Analysis 4: Comparison: Placebo vs PF-04937319 100 mg; [analysis description as in outcome 3, analysis 2]; Test type: Superiority or Other; p = 0.5066, t-test, 2 sided — P-value was 2-sided; LS Mean Difference = 0.30, 80% CI 2-sided [-0.28 to 0.88], Standard Error of Mean 0.452
Statistical Analysis 5: Comparison: Placebo vs Sitagliptin 100 mg; [analysis description as in outcome 3, analysis 2]; Test type: Superiority or Other; p = 0.8947, t-test, 2 sided — P-value was 2-sided; LS Mean Difference = -0.06, 80% CI 2-sided [-0.64 to 0.52], Standard Error of Mean 0.449
Statistical Analysis 6: Comparison: Placebo vs PF-04937319 3 mg; [analysis description as in outcome 2, analysis 5]; Test type: Superiority or Other; p = 0.0577, t-test, 2 sided — P-value was 2-sided; LS Mean Difference = 0.91, 80% CI 2-sided [0.30 to 1.52], Standard Error of Mean 0.478
Statistical Analysis 7: Comparison: Placebo vs PF-04937319 20 mg; [analysis description as in outcome 2, analysis 5]; Test type: Superiority or Other; p = 0.3012, t-test, 2 sided — P-value was 2-sided; LS Mean Difference = 0.51, 80% CI 2-sided [-0.12 to 1.14], Standard Error of Mean 0.490
Statistical Analysis 8: Comparison: Placebo vs PF-04937319 50 mg; [analysis description as in outcome 2, analysis 5]; Test type: Superiority or Other; p = 0.3165, t-test, 2 sided — P-value was 2-sided; LS Mean Difference = 0.48, 80% CI 2-sided [-0.13 to 1.09], Standard Error of Mean 0.476
Statistical Analysis 9: Comparison: Placebo vs PF-04937319 100 mg; [analysis description as in outcome 2, analysis 5]; Test type: Superiority or Other; p = 0.5191, t-test, 2 sided — P-value was 2-sided; LS Mean Difference = 0.31, 80% CI 2-sided [-0.31 to 0.93], Standard Error of Mean 0.481
Statistical Analysis 10: Comparison: Placebo vs Sitagliptin 100 mg; [analysis description as in outcome 2, analysis 5]; Test type: Superiority or Other; p = 0.5107, t-test, 2 sided — P-value was 2-sided; LS Mean Difference = 0.32, 80% CI 2-sided [-0.30 to 0.93], Standard Error of Mean 0.479
Statistical Analysis 11: Comparison: Placebo vs PF-04937319 3 mg; [analysis description as in outcome 2, analysis 6]; Test type: Superiority or Other; p = 0.1054, t-test, 2 sided — P-value was 2-sided; LS Mean Difference = 0.79, 80% CI 2-sided [0.17 to 1.42], Standard Error of Mean 0.488
Statistical Analysis 12: Comparison: Placebo vs PF-04937319 20 mg; [analysis description as in outcome 2, analysis 6]; Test type: Superiority or Other; p = 0.5341, t-test, 2 sided — P-value was 2-sided; LS Mean Difference = 0.31, 80% CI 2-sided [-0.33 to 0.96], Standard Error of Mean 0.502
Statistical Analysis 13: Comparison: Placebo vs PF-04937319 50 mg; [analysis description as in outcome 2, analysis 6]; Test type: Superiority or Other; p = 0.2782, t-test, 2 sided — P-value was 2-sided; LS Mean Difference = 0.53, 80% CI 2-sided [-0.10 to 1.15], Standard Error of Mean 0.487
Statistical Analysis 14: Comparison: Placebo vs PF-04937319 100 mg; [analysis description as in outcome 2, analysis 6]; Test type: Superiority or Other; p = 0.5331, t-test, 2 sided — P-value was 2-sided; LS Mean Difference = 0.31, 80% CI 2-sided [-0.32 to 0.94], Standard Error of Mean 0.492
Statistical Analysis 15: Comparison: Placebo vs Sitagliptin 100 mg; [analysis description as in outcome 2, analysis 6]; Test type: Superiority or Other; p = 0.9070, t-test, 2 sided — P-value was 2-sided; LS Mean Difference = 0.06, 80% CI 2-sided [-0.57 to 0.68], Standard Error of Mean 0.489
Statistical Analysis 16: Comparison: Placebo vs PF-04937319 3 mg; [analysis description as in outcome 3, analysis 16]; Test type: Superiority or Other; p = 0.1757, t-test, 2 sided — P-value was 2-sided; LS Mean Difference = 0.69, 80% CI 2-sided [0.04 to 1.35], Standard Error of Mean 0.512
Statistical Analysis 17: Comparison: Placebo vs PF-04937319 20 mg; [analysis description as in outcome 3, analysis 16]; Test type: Superiority or Other; p = 0.4083, t-test, 2 sided — P-value was 2-sided; LS Mean Difference = 0.44, 80% CI 2-sided [-0.24 to 1.11], Standard Error of Mean 0.527
Statistical Analysis 18: Comparison: Placebo vs PF-04937319 50 mg; [analysis description as in outcome 3, analysis 16]; Test type: Superiority or Other; p = 0.3150, t-test, 2 sided — P-value was 2-sided; LS Mean Difference = 0.51, 80% CI 2-sided [-0.14 to 1.17], Standard Error of Mean 0.511
Statistical Analysis 19: Comparison: Placebo vs PF-04937319 100 mg; [analysis description as in outcome 3, analysis 16]; Test type: Superiority or Other; p = 0.6631, t-test, 2 sided — P-value was 2-sided; LS Mean Difference = 0.23, 80% CI 2-sided [-0.44 to 0.89], Standard Error of Mean 0.516
Statistical Analysis 20: Comparison: Placebo vs Sitagliptin 100 mg; [analysis description as in outcome 3, analysis 16]; Test type: Superiority or Other; p = 0.8694, t-test, 2 sided — P-value was 2-sided; LS Mean Difference = -0.08, 80% CI 2-sided [-0.74 to 0.57], Standard Error of Mean 0.512
Statistical Analysis 21: Comparison: Placebo vs PF-04937319 3 mg; [analysis description as in outcome 3, analysis 21]; Test type: Superiority or Other; p = 0.2031, t-test, 2 sided — P-value was 2-sided; LS Mean Difference = 0.70, 80% CI 2-sided [0.00 to 1.40], Standard Error of Mean 0.545
Statistical Analysis 22: Comparison: Placebo vs PF-04937319 20 mg; [analysis description as in outcome 3, analysis 21]; Test type: Superiority or Other; p = 0.7137, t-test, 2 sided — P-value was 2-sided; LS Mean Difference = 0.21, 80% CI 2-sided [-0.52 to 0.93], Standard Error of Mean 0.563
Statistical Analysis 23: Comparison: Placebo vs PF-04937319 50 mg; [analysis description as in outcome 3, analysis 21]; Test type: Superiority or Other; p = 0.6810, t-test, 2 sided — P-value was 2-sided; LS Mean Difference = 0.22, 80% CI 2-sided [-0.48 to 0.92], Standard Error of Mean 0.545
Statistical Analysis 24: Comparison: Placebo vs PF-04937319 100 mg; [analysis description as in outcome 3, analysis 21]; Test type: Superiority or Other; p = 0.6921, t-test, 2 sided — P-value was 2-sided; LS Mean Difference = -0.22, 80% CI 2-sided [-0.92 to 0.49], Standard Error of Mean 0.550
Statistical Analysis 25: Comparison: Placebo vs PF-04937319 100 mg; Week 14 (Follow-up): Treatment difference and 80% CI were based on LS mean. MMRM analysis was performed with treatment, time and treatment-by-time interaction as fixed effects, baseline as the covariate, time was repeated for participant; Test type: Superiority or Other; p = 0.3702, t-test, 2 sided — P-value was 2-sided; LS Mean difference = -0.49, 80% CI 2-sided [-1.19 to 0.21], Standard Error of Mean 0.545

11. Secondary Outcome: Number of Participants With Abnormal Laboratory Values
Description: Hemoglobin,hematocrit,red blood cells(RBC) count:less than [<]0.8*lower limit of normal[LLN],platelets:<0.5*LLN/greater than [>]1.75*upper limit of normal [ULN],white blood cells(WBC):<0.6*LLN or >1.5*ULN,lymphocytes,total neutrophils:<0.8*LLN or >1.2*ULN, basophils,eosinophil,monocytes:>1.2*ULN;aspartate aminotransferase,alanine aminotransferase, alkaline phosphatase:>0.3*ULN,total protein,albumin:<0.8*LLN or >1.2*ULN;total bilirubin,direct bilirubin,indirect bilirubin:>1.5*ULN;triglycerides,cholesterol:>1.3*ULN, HDL:<0.8*LLN, LDL:>1.2*ULN,blood urea nitrogen,creatinine:>1.3*ULN,uric acid:>1.2*ULN;sodium: <0.95*LLN or >1.05*ULN,potassium,chloride,calcium,bicarbonate:<0.9*LLN or >1.1*ULN;creatine kinase:>2.0*ULN;glucose:<0.6*LLN or >1.5*ULN,urine WBC and RBC:>= 20/High Power Field [HPF]),urine epithelial cells (>=1 HPF),urine bacteria >20 high-powered field;qualitative urine glucose,urine blood to Hgb ratio (>=1);urine(protein,nitrite,mucus,leukocyte >=1 in urine dipstick test).
Time Frame: Baseline (Day 1) up to Week 14
Population: as for outcome 5
Measure: Number; unit: participants
Arm/Group | Placebo | PF-04937319 3 mg | PF-04937319 20 mg | PF-04937319 50 mg | PF-04937319 100 mg | Sitagliptin 100 mg
Number analyzed (Participants) | 56 | 57 | 53 | 56 | 55 | 55
participants | 46 | 49 | 45 | 46 | 53 | 43

ADVERSE EVENTS:
Description: Same event may appear as both AE and SAE. However, what is presented are distinct events. An event may be categorized as serious in 1 subject and nonserious in another subject, or 1 subject may have experienced both serious and nonserious event during study. AEs were also collected during the course of run-in period (metformin background therapy).
Arm/Group | Metformin 500 mg | Placebo | PF-04937319 3 mg | PF-04937319 20 mg | PF-04937319 50 mg | PF-04937319 100 mg | Sitagliptin 100 mg
Serious Adverse Events (participants affected / at risk) | 0/376 | 1/57 | 0/57 | 1/54 | 0/56 | 1/56 | 0/55
Other Adverse Events (participants affected / at risk) | 37/376 | 19/57 | 19/57 | 19/54 | 16/56 | 24/56 | 18/55
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Metformin 500 mg (N=376) | Placebo (N=57) | PF-04937319 3 mg (N=57) | PF-04937319 20 mg (N=54) | PF-04937319 50 mg (N=56) | PF-04937319 100 mg (N=56) | Sitagliptin 100 mg (N=55)
Myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Anal abscess (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Meningitis viral (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Metformin 500 mg (N=376) | Placebo (N=57) | PF-04937319 3 mg (N=57) | PF-04937319 20 mg (N=54) | PF-04937319 50 mg (N=56) | PF-04937319 100 mg (N=56) | Sitagliptin 100 mg (N=55)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 1 | 1 | 0
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Leukocytosis (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Bundle branch block right (Cardiac disorders) | 1 | 0 | 0 | 3 | 0 | 0 | 0
Type IIb hyperlipidaemia (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Type IV hyperlipidaemia (Congenital, familial and genetic disorders) | 3 | 1 | 1 | 0 | 1 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Hypothyroidism (Endocrine disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dry eye (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Eye inflammation (Eye disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Enteritis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Faeces discoloured (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Toothache (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 1 | 1 | 0
Vomiting (Gastrointestinal disorders) | 2 | 1 | 0 | 1 | 0 | 1 | 0
Asthenia (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Malaise (General disorders) | 2 | 0 | 1 | 1 | 0 | 0 | 0
Pain (General disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hepatitis (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Abscess neck (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Acute sinusitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Anal abscess (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Asymptomatic bacteriuria (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Body tinea (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Bronchitis (Infections and infestations) | 1 | 0 | 1 | 0 | 1 | 0 | 0
Conjunctivitis bacterial (Infections and infestations) | 1 | 0 | 1 | 0 | 0 | 0 | 0
Folliculitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 1 | 1 | 0 | 1 | 0 | 0 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Gingivitis (Infections and infestations) | 1 | 0 | 0 | 0 | 1 | 0 | 0
Helicobacter infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Influenza (Infections and infestations) | 1 | 0 | 0 | 2 | 0 | 2 | 0
Laryngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Malaria (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Mastitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 0 | 1 | 0 | 0 | 1 | 1 | 0
Osteomyelitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Otitis externa (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Otitis media (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Paronychia (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pharyngitis (Infections and infestations) | 3 | 0 | 0 | 0 | 0 | 0 | 0
Pyelonephritis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Respiratory tract infection viral (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 1 | 0
Subcutaneous abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Tonsillitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Tooth abscess (Infections and infestations) | 1 | 0 | 0 | 0 | 1 | 0 | 0
Tooth infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 2 | 1 | 1 | 4 | 0 | 1
Urinary tract infection (Infections and infestations) | 2 | 1 | 1 | 0 | 2 | 1 | 1
Viral infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Viral upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Muscle strain (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Blood pressure increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Blood triglycerides increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 1 | 0
Electrocardiogram ST segment elevation (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Haemoglobin decreased (Investigations) | 0 | 2 | 1 | 0 | 0 | 1 | 1
Hepatic enzyme increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Platelet count increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Vitamin B12 decreased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Weight decreased (Investigations) | 1 | 0 | 0 | 0 | 0 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 2 | 0 | 0 | 2 | 1 | 0 | 0
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 2 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 2 | 0 | 0 | 0 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0 | 1 | 0 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 1 | 0 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1 | 0 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0
Diabetic neuropathy (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 3 | 0 | 0 | 2 | 0 | 0 | 0
Facial paresis (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 2
Migraine (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0
Polyneuropathy (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Sciatica (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Syncope (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1
Nephropathy (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 2 | 2 | 1
Polyuria (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Proteinuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0
Pyuria (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Erectile dysfunction (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0 | 0 | 0 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 1 | 0 | 0 | 0 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Eczema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Psoriasis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 1 | 2 | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.